CLINICAL TRIAL: NCT05669443
Title: Application of Individualized Positive End-expiratory Pressure Using Electrical Impedance Tomography (EIT) in Patients Undergoing Robot Assisted Laparoscopic Prostatectomy : a Randomized Controlled Study
Brief Title: Effect of Optimized PEEP on Mechanical Ventilation During Robot Assisted Laparoscopic Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Chul Ho Chang, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 3-2022-0361
Record Dates: First submitted 2022-12-09; First posted 2022-12-30 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional PEEP (Experimental): Apply of PEEP 5
  Interventions: Device: conventional PEEP
- optimized PEEP (Active Comparator): Apply of optimized PEEP derived using EIT (airtom®)
  Interventions: Device: optimized PEEP

INTERVENTIONS:
Device: conventional PEEP — Maintain positive end expiratory pressure at 5 cmH2O throughout the surgery.
  Arms: conventional PEEP
Device: optimized PEEP — Immediately after induction of anesthesia, the patient remains unapplied to PEEP. After pneumoperitoneum + Trendelenburg posture, an appropriate PEEP value is derived using electrical impedance tomography (airtom®). And then derived value ( = optimized PEEP value) is applied until the end of the operation.
  Arms: optimized PEEP

SUMMARY:
Steep trendelenburg posture or pneumoperitoneum for surgery causes ventilation problems during surgery, so finding a way to overcome is a challenging task for anesthesiologists. In this study, for patients undergoing robot assisted laparoscopic prostatectomy under general anesthesia, anesthesia is going to perform by applying conventional positive end-expiratory pressure (PEEP 5cmH2O) or individually determined positive end-expiratory pressure values for each patient using electrical impedance tomography. We plan to compare intraoperative ventilation through arterial blood gas analysis to find out the way to improve intraoperative ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. 20 - 70 years of age who are scheduled for robotic assisted laparoscopic prostatectomy at the Department of Urology, Gangnam Severance Hospital,
2. ASA-PS (American Society of Anesthesiology Body Rating) I-IlI,
3. Patients with a BMI of 35 kg/m2 or less

Exclusion Criteria:

1. Patients with lung disease
2. BMI >35kg/m2
3. Patients for whom positive end-tidal pressure cannot be applied (large bullae, severe cardiac disease)
4. patient refusal

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 | end of surgery (before extubation)
  PaO2/FiO2 is the ratio of arterial oxygen partial pressure (PaO2) to oxygen fraction (FiO2), and is a commonly used indicator for evaluating pulmonary ventilation and diagnosing lung damage. Using this index, it is possible to determine whether oxygen obtained through the lungs is well delivered to the blood or not. It can be easily obtained by arterial blood gas analysis without complicated formulas or graphs.

SECONDARY OUTCOMES:
PaO2/FiO2 | 15 minutes after intubation, 1 hour after pnemoperitoneum
  partial pressure (PaO2) to oxygen fraction (FiO2), and is a commonly used indicator for evaluating pulmonary ventilation and diagnosing lung damage. Using this index, it is possible to determine whether oxygen obtained through the lungs is well delivered to the blood or not. It can be easily obtained by arterial blood gas analysis without complicated formulas or graphs.
ROI (region of interests) | 15 minutes after intubation, 1 hour after pnemoperitoneum, end of surgery (before extubation)
  region of interest using EIT
inhomogeneity index | 15 minutes after intubation, 1 hour after pnemoperitoneum, end of surgery (before extubation)
  inhomogeneity index : this index calculated from tidal EIT images representing the difference in impedance between the end of inspiration and the end of expiration.
total amount of fluid administered during surgery | end or surgery
total dose of vasopressor administered during surgery | end of surgery
length of hospitalization after surgery | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severacne Hospital Yonsei University College of Medicine, Seoul, South Korea